CLINICAL TRIAL: NCT02333201
Title: DYsphAgia In Mechanically Ventilated ICU patientS (DYnAMICS) - a Prospective Multicentre Observational Analysis
Brief Title: DYsphAgia In Mechanically Ventilated ICU patientS
Acronym: DYnAMICS
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Nestec S.A., Switzerland (Funding) (Unknown)
Responsible Party: Principal Investigator, Jörg Schefold, Principal Investigator/ Coordinating Investigator, Insel Gruppe AG, University Hospital Bern
Other Study IDs: Dynamics
Record Dates: First submitted 2014-12-22; First posted 2015-01-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Deglutition Disorders
Keywords: Deglutition Disorders; Dysphagia; Mechanical Ventilation; Sepsis
MeSH Terms: conditions — Deglutition Disorders; Sepsis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Dysphagia significantly contributes to morbidity and mortality in non-critically ill patients (as e.g. in stroke). Long term consequences of dysphagia include, among others, malnutrition, prolonged enteral tube feeding and increased risk of aspiration. In the present observational analysis, the investigators aim to elucidate the incidence and the impact of dysphagia on the clinical course of a mixed population of ICU patients post invasive mechanical ventilation.

DETAILED DESCRIPTION:
Dysphagia significantly contributes to morbidity and mortality in non-critically ill patients (as e.g. in stroke). Long term consequences of dysphagia include, among others, malnutrition, prolonged enteral tube feeding and increased risk of aspiration. In the present observational analysis, we aim to elucidate the incidence and the impact of dysphagia on the clinical course of a mixed population of ICU patients post invasive mechanical ventilation.

ICU patients are at increased risk for oropharyngeal dysphagia following endotracheal intubation. However, the incidence, respective underlying causes and clinical consequences of dysphagia in ICU patients are currently understudied. The impact on clinical outcomes of respective ICU patients thus remains currently unclear. A systematic review [1] reported highly variable dysphagia frequency rates depending on the time of mechanical ventilation/ intubation.

However, previous clinical trials were heterogeneous in design, methods of screening, and study outcome. The overall quality of evidence is considered low. The systematic review highlights the limited available evidence for dysphagia following intubation and hence the need for high-quality prospective trials. A recent retrospective single-centre trial [2] in a tertiary care ICU demonstrated a high presence of dysphagia in mechanical ventilated (MV) patients following extubation. Screening was performed using bedside swallowing evaluation (BSE).

In a prospective observational analysis, we aim to further elucidate the impact of dysphagia on respective clinical outcomes in ICU patients after mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria: all adult ICU patients post mechanical ventilation (observational analysis)

Exclusion Criteria:

* patients prone to die / moribund patients/ or dying patients
* patients post oesophageal resection / with oesophageal rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mixed Population of adult ICU patients (aged 18+) post invasive mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with dysphagia at discharge from ICU | expected average time frame about 72hrs. (at end of ICU stay/ discharge)

SECONDARY OUTCOMES:
Number of patients with dysphagia and dysphagia severity at first assessment | expected average time frame about 48 hrs.
Number of patients with dysphagia / incl. dysphagia severity at discharge | expected average time frame about 72 hrs. (end of ICU stay)
Number of patients with dysphagia in predefined patient categories: ICU-acquired weakness, stroke/ cerebrovascular infarction, traumatic brain injury, movement disorders, sepsis, cardiogenic, post abdominal surgery, trauma | during ICU stay (expected average length of ICU stay is about 72 hrs.)
Number of patients with dysphagia and (association to) sedatives prescribed | during ICU stay (expected average length of ICU stay is about 72 hrs.)
Number of patients re-intubated, reason for re-intubation, and antibiotic use | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period)
Number of patients with dysphagia and association to duration of mechanical ventilation | during ICU stay (expected average length of ICU stay is about 72 hrs.)
Number of patients with dysphagia (in association) to tube size, body weight/ BMI etc. | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period)
Number of patients with dysphagia according to disease severity and routine laboratory indices | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period)
Duration of dysphagia/ course of dysphagia severity during ICU/ hospital stay | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period, expected average length of hospital stay is about 14 days)
Number of chest X-ray examinations performed among patients w/ and w/o dysphagia | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period, expected average length of hospital stay is about 14 days)
Association of dysphagia and related ICU length of stay/ hospital length of stay | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period)
Association of dysphagia and related ICU- and intrahospital mortality/ readmission rate | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period)
Other clinical/ epidemiological factors associated with dysphagia (incl. descriptive analyses) | during ICU stay (expected average length of ICU stay is about 72 hrs./ observational period)

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Takala, Prof Dr., Study Chair — University of Bern, Inselspital; Stephan Jakob, Prof. Dr., Study Chair — University of Bern, Inselspital; Joerg C Schefold, MD, Principal Investigator — University of Bern, Inselspital
Locations (1):
- Dept. of Intensive Care Medicine, University of Bern,, Bern, Switzerland

REFERENCES:
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948
- [Background] Macht M, King CJ, Wimbish T, Clark BJ, Benson AB, Burnham EL, Williams A, Moss M. Post-extubation dysphagia is associated with longer hospitalization in survivors of critical illness with neurologic impairment. Crit Care. 2013 Jun 20;17(3):R119. doi: 10.1186/cc12791. PMID 23786755
- [Derived] Zuercher P, Schenk NV, Moret C, Berger D, Abegglen R, Schefold JC. Risk Factors for Dysphagia in ICU Patients After Invasive Mechanical Ventilation. Chest. 2020 Nov;158(5):1983-1991. doi: 10.1016/j.chest.2020.05.576. Epub 2020 Jun 7. PMID 32525018